CLINICAL TRIAL: NCT06688110
Title: Evaluation of Gixam's Efficacy Predicting Pre-cancerous Colorectal Polyps and Colorectal Cancer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jubaan Ltd. (Industry)
Collaborators: Jubaan GmbH (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Screening
Other Study IDs: CL-1004
Record Dates: First submitted 2024-11-12; First posted 2024-11-14 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Colorectal Cancer; Colorectal Adenomatous Polyp; Colorectal Neoplasms
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Colonoscopy

STUDY DESIGN:
Intervention Model Description: All enrolled subjects will undergo the Gixam test followed by a standard of care colonoscopy
Masking Description: Participants and physician performing colonoscopy will be blinded to the Gixam outcome
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Gixam followed by standard of care colonoscopy (Experimental): All enrolled participants will undergo the Gixam test followed by a standard of care colonoscopy
  Interventions: Device: Gixam System

INTERVENTIONS:
Device: Gixam System — Jubaan's Gixam System is designed to predict the likelihood of colorectal adenomas or SSL by using white light in the 400 to 720 nm range to capture ultra-high-definition images of the of the tongue and analyzing the spectral signature of the oral microbiome to predict the presence of colorectal adenomas or SSL with help of artificial intelligence (AI).
  Other Names: Colonoscopy

SUMMARY:
This is a prospective, single arm, multi-center clinical investigation aim to demonstrate the efficacy of Gixam in predicting the presence of premalignant colorectal polyps and colorectal cancer (CRC) in a fecal immunochemical test (FIT) positive population.

DETAILED DESCRIPTION:
1. Average risk persons eligible for CRC screening that have received a positive FIT outcome in the past 6 months and are scheduled for a screening colonoscopy at one of the participating centers will be offered to participate in the study.
2. Following the informed consent process, subjects will undergo the Gixam test.

   1. A subset of 50 subjects will participate in the repeatability assessment. They will undergo three (3) repetitive Gixam tests one after the other, by the same operator.
   2. Both the subject and the endoscopist will be blinded to the Gixam outcome
3. All subjects will thereafter undergo a standard of care HD-WL colonoscopy procedure.
4. All resected and retrieved lesions will be sent separately for histopathological evaluation.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects aged ≥50 - ≤80 years.
2. Able to provide a signed informed consent.
3. Underwent FIT screening within the past 6 months with a positive result.
4. Scheduled for a FIT positive screening colonoscopy at investigational site.

Exclusion Criteria:

1. Has undergone colonoscopy within the past nine (9) years, except for a failed colonoscopy due to poor bowel preparation, which must have been performed within the past year without therapeutic intervention.
2. Personal history of CRC.
3. Family history of CRC, defined as having one or more first-degree relatives (parent, sibling, or child) with CRC at any age.
4. Subject has a diagnosis or medical / family history of any of the following conditions, including:

   * Familial adenomatous polyposis (also referred to as "FAP", including attenuated FAP and Gardner's syndrome),
   * Hereditary non-polyposis CRC syndrome (also referred to as "HNPCC" or "Lynch Syndrome"),
   * Other hereditary cancer syndromes including but are not limited to Peutz-Jeghers Syndrome, MYH-Associated Polyposis (MAP), Turcot's (or Crail's) Syndrome, Cowden's Syndrome, Juvenile Polyposis, Neurofibromatosis, or Familial Hyperplastic Polyposis.
5. Subject has a diagnosis or personal history of inflammatory bowel disease (IBD) including chronic ulcerative colitis, and/or Crohn's disease, and/or IBD-undefined.
6. Subjects with the disability to extend their tongue.
7. Subjects with tongue piercing.
8. Dental visit in the 7 days prior to the Gixam test.
9. Intake of pro-biotics over the past 3 months pre-Gixam test.
10. Subject has any condition that in the opinion of the Investigator should preclude participation in the study.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Safety - number of device related adverse events and serious adverse events | Through study completion, up to 30 days
  Number of device related adverse events and serious adverse events
Efficacy - Gixam's sensitivity and specificity | Through study completion, up to 30 days
  Gixam's sensitivity and specificity to predict the presence of premalignant neoplastic colorectal polyps (advanced premalignant neoplastic lesions/non-advanced premalignant neoplastic lesion) and CRC

CONTACTS AND LOCATIONS:
Locations (1):
- Erasmus MC, Rotterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Jubaan's website — https://jubaan.com/